CLINICAL TRIAL: NCT01349244
Title: Correlation of Hydronephrosis on Point of Care Ultrasound With CT Finding in Patients With Expected Renal Colic
Brief Title: Hydronephrosis on Ultrasound With CT Finding in Patients With Renal Colic
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB # 1006006943
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Hydronephrosis; Renal Colic
Keywords: hydronephrosis; CT; POC US
MeSH Terms: conditions — Hydronephrosis; Renal Colic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the overall sensitivity and specificity of hydronephrosis on point-of-care bedside ultrasound to identify hydronephrosis as compared to hydronephrosis found by CT.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients 18 yrs or older with suspected renal colic in whom the clinician intends to obtain a CT scan to diagnose kidney stone.
* Informed consent will be required prior to enrollment in the study.

Exclusion Criteria:

* Known renal disease (any ESRD, transplant, PCKD), dementia, trauma, language barrier, incarcerated patients, and patients who do not undergo CT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective observational study involving a convenience sample of all ED patients scheduled for NCT at some point during their emergency department visit.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
hydronephrosis bedside ultrasound | Sept 2011-Jan 2013
  To determine the overall sensitivity and specificity of hydronephrosis on point-of-care bedside ultrasound to identify hydronephrosis as compared to hydronephrosis found on by CT.

SECONDARY OUTCOMES:
hydronephrosis bedside ultrasound | Sept 2011-Jan 2013
  To determine test performance characteristics of hydronephrosis on point of care ultrasound with the goal of incorporating POC US into a prospective rule for determining which patients with suspected renal colic require CT evaluation.

OTHER OUTCOMES:
hydronephrosis | Sept 2011-Jan 2013
  To prospectively correlate the finding and degree of hydronephrosis on point of care ultrasound with stone size (a marker for likely spontaneous passage).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Moore, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, Emergency Department, New Haven, Connecticut, United States